CLINICAL TRIAL: NCT00383266
Title: A Phase II Study of Pemetrexed and Carboplatin in the Treatment of Esophageal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0541 / 201103198
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed + Carboplatin (Experimental): * Pemetrexed 500 mg/m^2 IV over 10 minutes
  * Carboplatin AUC 5 IV over 30 minutes on day 1 of each cycle
  * Each cycle will last 21 days.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Pemetrexed
Drug: Carboplatin

SUMMARY:
This is a study of an investigational agent, pemetrexed, in combination with a standard chemotherapy drug, carboplatin, for treatment of patients with metastatic esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically proven metastatic or recurrent esophageal cancer. Both adenocarcinoma and squamous carcinoma are eligible for the study. Patients with small cell carcinoma or sarcoma of the esophagus are not eligible for the study.
* Patients may have had no prior chemotherapy treatment for metastatic esophageal cancer. Patients may have had chemotherapy with 5-FU combined with definitive radiotherapy for curative intent in the adjuvant, neoadjuvant, or definite setting for locally advanced esophageal cancer, if no less than one year prior to trial enrollment. Patients may not have received pemetrexed in the past.
* Patients who have had radiotherapy for esophageal cancer must have completed radiotherapy at least four weeks prior to entry in the study.
* Patients need to have measurable disease.
* Lesions that are not considered measurable include the following:

  * Bone lesions
  * Brain metastases or leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
  * Tumor lesions situated in a previously irradiated area
* ECOG) performance status of 0-2.
* Life expectancy of >=12 weeks.
* Patients must have adequate bone marrow function defined as: white blood cells (WBC) >= 3000/mm^3, absolute neutrophil count (ANC) >= 1,500/mm^3, hemoglobin >= 9.0 g/dL, and platelet count >= 100,000/mm^3.
* Patients must have adequate liver function defined as: Bilirubin <= 1.5 x institutional normal and ALT/AST < 3 x institutional normal.
* Patients must have adequate renal function defined as: serum creatinine <= 3.0 mg/dL and creatinine clearance >= 45 mL/min.
* Radiation therapy for brain metastases should be completed at least four weeks prior to enrollment to this protocol.
* Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or uncontrolled symptomatic cardiac arrhythmia.
* Patients must be able to be compliant with premedications of dexamethasone, folic acid, and vitamin B12.
* For all sexually active women of child-bearing age, the use of adequate contraception (hormonal or barrier method of birth control) will be required prior to study entry and for the duration of study participation.
* Age >= 18 years.

  * Written consent.
  * Ibuprofen (400 mg qid) can be administered with Alimta in patients with normal renal function (creatinine clearance > 80 mL/min

Exclusion Criteria:

* Patients with third-space fluid (pleural effusions, ascites, etc.) uncontrolled by drainage.
* Pregnant or nursing females
* Patients who have had pre-existing neuropathy greater than or equal to grade 2.
* Patients with known active CNS metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Q. Baggstrom, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 10/11/2006 and closed to participant enrollment on 11/12/2009.
Period: Overall Study
Arm/Group | Pemetrexed + Carboplatin
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed + Carboplatin: * Pemetrexed 500 mg/m2 IV over 10 minutes
  * Carboplatin AUC 5 IV over 30 minutes on day 1 of each cycle
  * Each cycle will last 21 days.
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: * Overall response rate = complete response (CR) + partial response (PR) using RECIST.
  * CR=disappearance of all target lesions and disappearance of all non-target lesions and normalization of tumor marker level
  * PR=at least a 30% decrease in the sum of the longest diameter (LD) of the target lesions taking as reference the baseline sum LD
Time Frame: Until patient progresses or dies (median follow-up 293 days -- range (63-632 days)
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 9
percentage of participants
  Complete response | 0
  Partial response | 33

2. Secondary Outcome: Time to Disease Progression
Description: -Progressive disease=at least a 20% increase in the sum of the LD of the target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: Until patient progresses (median follow-up 293 days -- range (63-632 days)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 9
months | 3.6 [1.1 to 7.4]

3. Secondary Outcome: Overall Survival Rate
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 9
percentage of participants | 22.2

4. Secondary Outcome: Toxicities
Time Frame: 30 days following completion of treatment (maximum number of cycles = 6)
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 9
participants
  Cardiac ischemia/infarction | 1
  Pancreatitis | 1
  Tumor pain | 1
  Chest/thorax pain | 1
  Hemoglobin | 8
  Chest pain | 1
  Dry eye syndrome | 1
  Abdominal pain | 2
  Constipation | 3
  Diarrhea | 3
  Dysphagia | 1
  Hiccoughs | 1
  Mucositis | 2
  Nausea | 6
  Oral cavity pain | 1
  Stomatitis | 1
  Vomiting | 4
  Chills | 2
  Edema | 1
  Fatigue | 5
  Fever | 1
  Sweating | 5
  Colitis (c. difficile) | 1
  Infection without neutropenia | 1
  ALT | 4
  AST | 2
  Alkaline phosphtase | 2
  Leukocytes (WBC) | 3
  Low CO2 | 2
  Lymphopenia | 6
  Neutrophils | 2
  Platelets | 1
  Weight loss | 1
  Anorexia | 2
  Dehydration | 1
  Hypercalcemia | 1
  Hyperglycemia | 3
  Hyperkalemia | 3
  Hypernatremia | 3
  Hypoalbuminemia | 3
  Hypocalcemia | 1
  Hypoglycemia | 1
  Hypokalemia | 1
  Hyponatremia | 1
  Lipase | 1
  Back pain | 1
  Hernia | 1
  Limb pain | 1
  Dizziness | 3
  Headache | 3
  Neuropathy - motor | 1
  Neuropathy - sensory | 5
  Insomnia | 4
  Mood alteration - anxiety | 2
  Creatinine | 1
  Creatinine clearance | 1
  Allergic rhintis | 2
  Cough | 4
  Dyspnea | 3
  Hemorrhage - nose | 1
  Alopecia | 1
  Dry skin | 2
  Other: skin | 1
  Puritis | 1
  Rash | 1
  Skin breakdown/decubitous ulcer | 1
  Hot flash | 1

5. Secondary Outcome: Overall Survival Rate
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 9
percentage of participants | 0

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from initiation of treatment to the date of any reason death while those living subjects will be censored at the last assessment date.
Time Frame: Until patient's death (median follow-up 293 days -- range (63-632 days))
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 9
months | 9.6 [2.1 to 17.5]

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Carboplatin
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed + Carboplatin (N=9)
Pancreatitis (Gastrointestinal disorders) | 1
Chest/thorax pain (Respiratory, thoracic and mediastinal disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed + Carboplatin (N=9)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Chills (General disorders) | 2
Edema (General disorders) | 1
Fatigue (General disorders) | 5
Fever (General disorders) | 1
Hot flash (Vascular disorders) | 1
Sweating (General disorders) | 5
Weight loss (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Skin breakdown/decubitous ulcer (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Other: skin (Skin and subcutaneous tissue disorders) | 1
Puritis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Hiccoughs (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 8
Leukocytes (WBC) (Investigations) | 3
Lymphopenia (Investigations) | 6
Neutrophils (ANC) (Investigations) | 2
Platelets (Investigations) | 1
Hemorrhage - nose (Respiratory, thoracic and mediastinal disorders) | 1
Infection without neutropenia (Infections and infestations) | 1
Colitis (c. difficile) (Infections and infestations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Alkaline phosphatase (Investigations) | 2
ALT (Investigations) | 4
AST (Investigations) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Low CO2 (Investigations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1
Lipase (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 4
Mood alteration - anxiety (Psychiatric disorders) | 2
Neuropathy - sensory (Nervous system disorders) | 5
Neuropathy - motor (Nervous system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chest pain (Cardiac disorders) | 1
Oral cavity pain (Gastrointestinal disorders) | 1
Limb pain (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine (Renal and urinary disorders) | 1
Creatinine clearance (Renal and urinary disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Hernia (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to lack of participant accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes